CLINICAL TRIAL: NCT06625736
Title: Anti-obesity Effects of Dandelion (Taraxacum Officinale L.) in Premenopausal Obese Women: Impacts on Appetite, Energy Intake and Lipid Metabolism
Brief Title: Anti-obesity Effects of Dandelion (Taraxacum Officinale L.)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: October 6 University (Other)
Collaborators: Pharos University in Alexandria (Other)
Responsible Party: Principal Investigator, rabab ahmed mohamed, Principle investigator, October 6 University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Dandelion effect on obesity
Record Dates: First submitted 2024-09-30; First posted 2024-10-03 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-09

CONDITIONS: Obese Women; Perimenopause
Keywords: Dandelion; Premenopausal Obese Women; Anti-obesity
MeSH Terms: interventions — Orlistat

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control group (Active Comparator): The Xenical group:60 patients will receive identical capsules of 120mg (one capsule) to be taken three times daily with meals and for 12 weeks, equaling 360mg total daily dose.
  Interventions: Drug: Xenical
- The dandelion extract group (Experimental): The dandelion extract group: 60 patients will receive 500 mg capsules of dandelion leaf extract, given 3 times per day before meals and for 12 weeks.
  Interventions: Dietary Supplement: The dandelion extract

INTERVENTIONS:
Drug: Xenical — The Xenical group will receive identical capsules 120mg (one capsule) to be taken three times daily with meals, equaling 360mg total daily dose, which aligns with the usage in adult female patients
  Arms: Control group
Dietary Supplement: The dandelion extract — The dandelion extract group will receive 500 mg capsules of dandelion leaf extract, given 3 times per day before meals.
  Arms: The dandelion extract group

SUMMARY:
The study investigates the effectiveness of the natural product Dandelion in treating obesity in premenopausal women through a randomized interventional trial, measuring various parameters and biomarkers.

DETAILED DESCRIPTION:
The study aims to explore the anti-obesity effects of dandelion supplementation in premenopausal obese women. The research will measure changes in appetite, energy intake, body weight, composition, lipid profile, and inflammatory markers, providing evidence of dandelion's efficacy as an anti-obesity phototherapy. The randomized interventional trial will measure multiple parameters and biomarkers.

ELIGIBILITY:
Inclusion Criteria:

Premenopausal women with obesity. Age between 18-45 years Stable body weight in the past 3 months

Exclusion Criteria:

Pregnancy Breastfeeding Diabetes Cardiovascular diseases kidney or liver diseases use of medications that affect body weight Smoking Allergy to dandelion or related plants

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Premenopausal Women
Enrollment: 120 (Actual)
Dates: Start 2024-01-05 (Actual); Primary Completion 2024-09-07 (Actual); Study Completion 2024-09-07 (Actual)

PRIMARY OUTCOMES:
Changes in body weight | monthly change, assessed up to 3 months
Change in fat mass | Monthly change, assessed up to 3 months

SECONDARY OUTCOMES:
Appetite Ratings | monthly change, assessed up to 3 months
Dietary intake via 24-hour recalls | Recorded for patients daily, assessed up to 3 months
Lipid profile | Monthly change, assessed up to 3 months
CRP | Monthly change, assessed up to 3 months
  C-reactive protein
TNF-α | Monthly change, assessed up to 3 months
IL-6 | Monthly change, assessed up to 3 months
  Interelukine 6
IL-16 | Monthly change, assessed up to 3 months
Glycemic indices | Monthly change, assessed up to 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- October 6 University Hospital, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided